CLINICAL TRIAL: NCT00197236
Title: Immunogenicity and Safety of GSK Biologicals' Inactivated Hepatitis A Vaccine (Havrix™) Co-administered With GSK Biologicals' DTaP Vaccine (Infanrix™) and Aventis Pasteur's Haemophilus b Conjugate Vaccine (ActHIB) in Healthy Children 15 Months of Age
Brief Title: Immunogenicity and Safety of Havrix™ Co-Administered With a Diphtheria, Tetanus and Pertussis and a Haemophilus b Vaccine in Children Aged 15 Months
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 208109/232
Record Dates: First submitted 2005-09-15; First posted 2005-09-20 (Estimated); Results first posted 2009-07-24 (Estimated); Last update posted 2018-08-20 (Actual); Status verified 2017-01

CONDITIONS: Hepatitis A
Keywords: Hepatitis A
MeSH Terms: conditions — Hepatitis A | interventions — Hepatitis A Vaccines; Diphtheria-Tetanus-acellular Pertussis Vaccines; Haemophilus influenza type b polysaccharide vaccine-tetanus toxin conjugate

ARMS (3):
- Havrix Group (Active Comparator): Subjects received one dose of Havrix at Day 0 followed by a second dose of Havrix at Month 6-9.
  Interventions: Biological: Havrix™
- Infanrix + ActHIB→Havrix Group (Experimental): Subjects received Infanrix co-administered with ActHIB at Day 0, followed by one dose of Havix at Day 30 and a second dose of Havrix at Month 7-10.
  Interventions: Biological: Havrix™; Biological: Infanrix™; Biological: ActHIB™
- Havrix + Infanrix + ActHIB Group (Active Comparator): Subjects received one dose of Havrix co-administered with Infanrix and ActHIB vaccines at Day 0 followed by a second dose of Havrix at Month 6-9.
  Interventions: Biological: Havrix™; Biological: Infanrix™; Biological: ActHIB™

INTERVENTIONS:
Biological: Havrix™ — 2 intramuscular injections, 6 months apart
Biological: Infanrix™ — 1 intramuscular injection
  Arms: Havrix + Infanrix + ActHIB Group; Infanrix + ActHIB→Havrix Group
Biological: ActHIB™ — 1 intramuscular injection
  Arms: Havrix + Infanrix + ActHIB Group; Infanrix + ActHIB→Havrix Group

SUMMARY:
This is a study to evaluate the immune response and safety of GSK Biologicals 2-dose inactivated hepatitis A vaccine when administered with a diphtheria, tetanus and pertussis combination (DTaP) vaccine and a Haemophilus influenza type B (Hib) vaccine in children 15 months of age. The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

DETAILED DESCRIPTION:
An open, controlled comparison of Havrix™ administered alone or with Infanrix™ and ActHIB. The three groups evaluated are: 1) Havrix™ alone, 2) Havrix™ + Infanrix™ and ActHIB and 3) Infanrix™ and ActHIB followed by Havrix™ one month later.

ELIGIBILITY:
Inclusion Criteria:

* Subjects whose parents/guardians are believed by the investigator to be willing to comply with the requirements of the protocol
* A male or female child 12 or 13 months of age at the time of entry into the Enrolment Phase,
* Subjects must have previously received three doses each of DTaP and Hib vaccines during the first year of life. The three doses of DTaP vaccine must have been administered as either Infanrix™ or Pediarix™ and the three doses of Hib vaccine must have been administered as ActHIB™, HibTITER™, OmniHIB™.
* Subjects who, at 15 months of age, will have had at least six months elapse since their third dose of Infanrix™ or Pediarix™,
* Written informed consent obtained from the parents or guardian of the subject,
* Free of obvious health problems as established by medical history and history-directed physical examination before entering into the study, and
* Parents/guardian of the subject must have a telephone or be able to be contacted by telephone.

Exclusion Criteria:

* Use of any investigational or non-registered drug or vaccine other than the study vaccine(s) within 31 days preceding the first dose of study vaccine, or planned use during the study period,
* Chronic administration (defined as more than 14 days) of immuno-suppressant or other immune-modifying drugs within six months prior to vaccination or planned administration at any time during the study period.
* Planned administration or administration of any vaccine not foreseen by the study protocol during the period 42 days before and 31 days after each dose of study vaccine(s).
* Previous vaccination against DTaP using a commercially-available brand other than Infanrix™ or Pediarix™ or against Hib using a commercially-available brand other than ActHIB™, HibTITER™ or OmniHIB™.
* Previous vaccination with more than three doses of DTaP-containing vaccines or more than three doses of Hib-containing vaccines.
* Previous vaccination against hepatitis A,
* History or known exposure to hepatitis A,
* History of diphtheria, tetanus, pertussis and/or Haemophilus influenza type b,
* Known exposure to diphtheria, tetanus, pertussis and/or Haemophilus influenza type b within 31 days prior to the start of the study,
* History of non-response to any vaccine in the current routine immunization schedule,
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection,
* A family history of congenital, hereditary or infectious immunodeficiency or parental risk factors for HIV infection,
* History of allergic disease/reactions or hypersensitivity likely to be exacerbated by any component of Havrix™, Infanrix™ or ActHIB™ including 2-phenoxyethanol, neomycin and gelatin,
* History of hypersensitivity/allergic reaction to latex
* Major congenital defects or serious chronic illness,
* History of any neurologic disorder
* Acute disease at the time of vaccination.
* Administration of immunoglobulins and/or any blood products within three months prior to the first dose of study vaccine or planned administration at any time during the entire study period, i.e., the Enrolment Phase, the Active Phase and the Extended Safety Follow-up Phase

Ages: 12 Months to 13 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 468 (Actual)
Dates: Start 2003-11-11; Primary Completion 2007-12-03 (Actual); Study Completion 2007-12-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (21):
- United States (21):
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Oakland, California
  - GSK Investigational Site, San Ramon, California
  - GSK Investigational Site, Wilmington, Delaware
  - GSK Investigational Site, Pembroke Pines, Florida
  - GSK Investigational Site, Martinez, Georgia
  - GSK Investigational Site, Waterloo, Iowa
  - GSK Investigational Site, Bossier City, Louisiana
  - GSK Investigational Site, Long Branch, New Jersey
  - GSK Investigational Site, Ithaca, New York
  - GSK Investigational Site, Bismarck, North Dakota
  - GSK Investigational Site, Youngstown, Ohio
  - GSK Investigational Site, Bellevue, Pennsylvania
  - GSK Investigational Site, Hershey, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Beaumont, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Danville, Virginia
  - GSK Investigational Site, Mechanicsville, Virginia
  - GSK Investigational Site, La Crosse, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Trofa AF, Klein NP, Paul IM, Michaels MG, Goessler M, Chandrasekaran V, Blatter M. Immunogenicity and safety of an inactivated hepatitis A vaccine when coadministered with Diphtheria-tetanus-acellular pertussis and haemophilus influenzae type B vaccines in children 15 months of age. Pediatr Infect Dis J. 2011 Sep;30(9):e164-9. doi: 10.1097/INF.0b013e31821b8a7d. PMID 21494175
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 208109/232 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 208109/232 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 208109/232 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 208109/232 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 208109/232 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 208109/232 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the total of 468 subjects enrolled, only 394 were vaccinated and as such considered as 'started'.
Period: Overall Study
Arm/Group | Havrix Group | Havrix + Infanrix + ActHIB Group | Infanrix + ActHIB→Havrix Group
Started | 135 | 127 | 132
Completed | 121 | 110 | 109
Not Completed | 14 | 17 | 23
Not completed — Adverse Event | 1 | 0 | 1
Not completed — Lost to Follow-up | 5 | 14 | 6
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Withdrawal by Subject | 7 | 3 | 11
Not completed — Study drug/medication expiration | 1 | 0 | 3
Not completed — Returned out of specified time window | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Havrix Group | Havrix + Infanrix + ActHIB Group | Infanrix + ActHIB→Havrix Group | Total
Number analyzed (Participants) | 135 | 127 | 132 | 394
Age, Continuous [Mean (Standard Deviation); unit: months] | 15.1 (0.36) | 15.1 (0.3) | 15.0 (0.21) | 15.1 (0.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 64 | 67 | 186
  Male | 80 | 63 | 65 | 208

OUTCOME MEASURES:

1. Primary Outcome: Number of Seropositive Subjects for Anti-hepatitis A Virus (HAV) Antibodies Following the Second Dose of Havrix
Description: Subjects are defined as being anti-HAV seropositive if their anti-HAV antibody concentration is ≥ 15 milli-International Units per milliliter (mIU/mL).
Time Frame: 31 days following the second dose of Havrix™
Population: Analysis was performed on the According-to-Protocol cohort for immunogenicity including subjects who had at least one study vaccine administered and for whom assay results were available for antibodies against at least one study vaccine antigen component after vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Havrix Group | Havrix + Infanrix + ActHIB Group | Infanrix + ActHIB→Havrix Group
Number analyzed (Participants) | 88 | 84 | 77
Participants | 88 | 84 | 77

2. Primary Outcome: Number of Anti-diphtheria, Anti-tetanus and Anti-polyribosylribitol Phosphate (PRP) Seroprotected Subjects
Description: Subjects are defined as being anti-diphtheria, anti-tetanus and anti-PRP seroprotected if their anti-diphtheria and anti-tetanus antibody concentration is ≥ 0.1 International Units per milliliter (IU/mL) and if their anti-PRP antibody concentration is ≥ 1 microgram per milliliter (μg/mL), respectively.
Time Frame: 31 days following the administration of Infanrix™ and ActHIB
Population: Analysis was performed on the According-to-Protocol cohort for immunogenicity, only for those groups receiving Infanrix and ActHIB vaccines.
Measure: Count of Participants; unit: Participants
Arm/Group | Havrix + Infanrix + ActHIB Group | Infanrix + ActHIB→Havrix Group | Havrix Group
Number analyzed (Participants) | 90 | 80 | 0
Participants
  Anti-diphtheria: number analyzed (Participants) | 89 | 80 | 0
  Anti-diphtheria | 89 | 80 |
  Anti-tetanus: number analyzed (Participants) | 88 | 80 | 0
  Anti-tetanus | 88 | 80 |
  Anti-PRP: number analyzed (Participants) | 90 | 79 | 0
  Anti-PRP | 90 | 77 |

3. Primary Outcome: Number of Vaccine Responders for Anti-pertussis Toxoid (PT), Anti-filamentous Hemagglutinin (FHA) and Anti-pertactin (PRN)
Description: Subjects are considered as being vaccine responders if they were initially seronegative and become seropositive (≥ 5 Enzyme Linked Immunosorbent Assay Units per Milliliter (EL.U/mL)), or were initially seropositive and have a 2-fold increase above pre-study concentrations.
Time Frame: 31 days following the administration of Infanrix™ and ActHIB
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Havrix + Infanrix + ActHIB Group | Infanrix + ActHIB→Havrix Group | Havrix Group
Number analyzed (Participants) | 88 | 76 | 0
Participants
  Anti-PT: number analyzed (Participants) | 88 | 74 | 0
  Anti-PT | 87 | 71 |
  Anti-FHA | 85 | 75 |
  Anti-PRN: number analyzed (Participants) | 88 | 75 | 0
  Anti-PRN | 86 | 74 |

4. Secondary Outcome: Anti-diphtheria and Anti-tetanus Antibody Geometric Mean Concentrations (GMC)
Description: GMCs are expressed as International Units per milliliter (IU/mL).
Time Frame: 31 days following the administration of Infanrix™ and ActHIB
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Havrix + Infanrix + ActHIB Group | Infanrix + ActHIB→Havrix Group | Havrix Group
Number analyzed (Participants) | 89 | 80 | 0
IU/mL
  Anti-diphtheria | 11.3 [9.8 to 13.1] | 10.3 [8.7 to 12.3] |
  Anti-tetanus: number analyzed (Participants) | 88 | 80 | 0
  Anti-tetanus | 7.0 [5.9 to 8.2] | 7.3 [6.0 to 8.8] |

5. Secondary Outcome: Anti-polyribosylribitol Phosphate (PRP) Antibody Geometric Mean Concentrations (GMC)
Description: GMCs are expressed as microgram/milliliter (µg/mL).
Time Frame: 31 days following the administration of Infanrix™ and ActHIB
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Havrix + Infanrix + ActHIB Group | Infanrix + ActHIB→Havrix Group | Havrix Group
Number analyzed (Participants) | 90 | 79 | 0
µg/mL | 60.8 [45.9 to 80.4] | 41.0 [30.0 to 55.9] |

6. Secondary Outcome: Number of Subjects Seropositive for Anti-pertussis Toxoid (PT), Anti-filamentous Hemagglutinin (FHA), Anti-pertactin (PRN) and Anti-polyribosylribitol Phosphate (PRP)
Description: Seropositivity is defined as antibody concentrations ≥ 5 Enzyme Linked Immunosorbent Assay Units per Milliliter (EL.U/mL) for anti-PT, anti-FHA and anti-PRN antibodies and as antibody concentrations ≥ 0.15 microgram/milliliter (µg/mL) for anti-PRP antibodies.
Time Frame: 31 days following the administration of Infanrix™ and ActHIB
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Havrix + Infanrix + ActHIB Group | Infanrix + ActHIB→Havrix Group | Havrix Group
Number analyzed (Participants) | 90 | 80 | 0
Participants
  Anti-PT: number analyzed (Participants) | 89 | 80 | 0
  Anti-PT | 89 | 80 |
  Anti-FHA: number analyzed (Participants) | 89 | 80 | 0
  Anti-FHA | 89 | 80 |
  Anti-PRN: number analyzed (Participants) | 89 | 80 | 0
  Anti-PRN | 89 | 80 |
  Anti-PRP: number analyzed (Participants) | 90 | 79 | 0
  Anti-PRP | 90 | 79 |

7. Secondary Outcome: Number of Seropositive Subjects for Anti-hepatitis A Virus (HAV) Antibodies Following the First Dose of Havrix
Description: as for outcome 1
Time Frame: 31 days following the first dose of Havrix™
Population: Analysis was performed on the According-to-Protocol cohort for immunogenicity, only for the Havrix Group and the Havrix + Infanrix + ActHIB Group.
Measure: Count of Participants; unit: Participants
Arm/Group | Havrix Group | Havrix + Infanrix + ActHIB Group | Infanrix + ActHIB→Havrix Group
Number analyzed (Participants) | 94 | 89 | 0
Participants | 82 | 77 |

8. Secondary Outcome: Anti-hepatitis A Virus (HAV) Antibody Geometric Mean Concentrations (GMC) Following the First Dose of Havrix
Description: Anti-hepatitis A (HAV) antibody geometric mean concentrations (GMC) are expressed as milli-International Units per milliliter (mIU/mL).
Time Frame: 31 days following the first dose of Havrix™
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Havrix Group | Havrix + Infanrix + ActHIB Group | Infanrix + ActHIB→Havrix Group
Number analyzed (Participants) | 94 | 89 | 0
mIU/mL | 51.5 [41.7 to 63.7] | 51.5 [41.8 to 63.5] |

9. Secondary Outcome: Anti-hepatitis Virus A (HAV) Antibody Geometric Mean Concentrations (GMC) Following the Second Dose of Havrix
Description: as for outcome 8
Time Frame: 31 days following the second dose of Havrix™
Population: Analysis was performed on the According-to-Protocol cohort for immunogenicity.
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Havrix Group | Havrix + Infanrix + ActHIB Group | Infanrix + ActHIB→Havrix Group
Number analyzed (Participants) | 88 | 84 | 77
mIU/mL | 1700.4 [1306.0 to 2213.7] | 1904.4 [1552.7 to 2335.7] | 1625.1 [1378.2 to 1916.3]

10. Secondary Outcome: Number of Subjects With Vaccine Response to Havrix™.
Description: Vaccine response to Havrix is defined as post-vaccination anti-HAV antibody concentrations ≥ 15 mIU/mL in initially seronegative subjects or a ≥ 2-fold increase above the pre-vaccination anti-HAV antibody concentration in initially seropositive subjects.
Time Frame: 31 days following the second dose
Population: Analysis was performed on the According-to-Protocol cohort for immunogenicity
Measure: Count of Participants; unit: Participants
Arm/Group | Havrix Group | Havrix + Infanrix + ActHIB Group | Infanrix + ActHIB→Havrix Group
Number analyzed (Participants) | 86 | 83 | 74
Participants | 86 | 83 | 74

11. Secondary Outcome: Number of Subjects Reporting Solicited Local Adverse Events (AEs)
Description: Solicited local AEs assessed include pain, redness and swelling. Data across doses are presented in the table.
Time Frame: 4-day period following each dose of study vaccine(s)
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Havrix Group | Havrix + Infanrix + ActHIB Group | Infanrix + ActHIB→Havrix Group
Number analyzed (Participants) | 130 | 118 | 122
Participants
  Pain | 44 | 60 | 70
  Redness | 34 | 54 | 63
  Swelling | 21 | 38 | 46

12. Secondary Outcome: Number of Subjects Reporting Solicited General Adverse Events (AEs)
Description: Solicited general AEs assessed include drowsiness, axillary fever ≥ 37.5°C, irritability and loss of appetite. Data across doses are presented in the table.
Time Frame: 4-day period following each dose of study vaccine(s)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Havrix Group | Havrix + Infanrix + ActHIB Group | Infanrix + ActHIB→Havrix Group
Number analyzed (Participants) | 130 | 118 | 123
Participants
  Drowsiness | 44 | 50 | 53
  Fever | 16 | 26 | 31
  Irritability | 56 | 62 | 70
  Loss of appetite | 33 | 40 | 48

13. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events (AEs)
Description: An Adverse Event is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: 31-day period following each dose of study vaccine(s)
Population: The analysis was performed on the Total Vaccinated Cohort
Measure: Count of Participants; unit: Participants
Arm/Group | Havrix Group | Havrix + Infanrix + ActHIB Group | Infanrix + ActHIB→Havrix Group
Number analyzed (Participants) | 135 | 127 | 132
Participants | 75 | 69 | 71

14. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs), New Chronic Illnesses and Medically Significant Events
Description: Since the related information about medically significant events was not specifically collected and new chronic illnesses were only collected in the extended safety follow-up phase, all unsolicited adverse events (AEs) throughout the study are reported in the table without identifying which event was a medically significant or new chronic illness.
Time Frame: Active Phase and the 6-months Extended Safety Follow-up (ESFU) Phase.
Population: The analyses were performed on the Total Vaccinated Cohort for the active phase of the study and on the Extended safety follow-up cohort for the 6-month extended follow-up (ESFU) phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Havrix Group | Havrix + Infanrix + ActHIB Group | Infanrix + ActHIB→Havrix Group
Number analyzed (Participants) | 135 | 127 | 132
Participants
  SAEs | 5 | 2 | 4
  AEs during Active Phase | 80 | 74 | 72
  AEs during ESFU: number analyzed (Participants) | 119 | 111 | 109
  AEs during ESFU | 11 | 10 | 7

ADVERSE EVENTS:
Arm/Group | Havrix Group | Havrix + Infanrix + ActHIB Group | Infanrix + ActHIB→Havrix Group
Serious Adverse Events (participants affected / at risk) | 5 | 2 | 4
Other Adverse Events (participants affected / at risk) | 95/135 | 105/127 | 107/132
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Havrix Group | Havrix + Infanrix + ActHIB Group | Infanrix + ActHIB→Havrix Group
Dehydration (Metabolism and nutrition disorders) | 2/135 | 0/127 | 1/132
Gastroenteritis (Infections and infestations) | 1/135 | 1/127 | 0/132
Developmental delay (General disorders) | 1/135 | 0/127 | 1/132
Expressive language disorder (Psychiatric disorders) | 1/135 | 0/127 | 1/132
Arthritis bacterial (Infections and infestations) | 1/135 | 0/127 | 0/132
Asthma (Respiratory, thoracic and mediastinal disorders) | 1/135 | 0/127 | 0/132
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0/135 | 0/127 | 1/132
Failure to thrive (Metabolism and nutrition disorders) | 1/135 | 0/127 | 0/132
Pyrexia (General disorders) | 0/135 | 1/127 | 0/132
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0/135 | 0/127 | 1/132
Tachycardia (Cardiac disorders) | 0/135 | 1/127 | 0/132
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0/135 | 0/127 | 1/132
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Havrix Group (N=135) | Havrix + Infanrix + ActHIB Group (N=127) | Infanrix + ActHIB→Havrix Group (N=132)
Diarrhea (Gastrointestinal disorders) | 9 | 4 | 7
Teething (Gastrointestinal disorders) | 3 | 8 | 4
Vomiting (Gastrointestinal disorders) | 7 | 4 | 4
Pyrexia (General disorders) | 9 | 7 | 9
Otitis media (Infections and infestations) | 13 | 11 | 22
Upper respiratory tract infection (Infections and infestations) | 18 | 18 | 16
Viral infection (Infections and infestations) | 3 | 7 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 4 | 14
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 5 | 4 | 14
Pain at the injection site (General disorders) | 44 | 60 | 70
Redness at the injection site (General disorders) | 34 | 54 | 63
Swelling at the injection site (General disorders) | 21 | 38 | 46
Drowsiness (General disorders) | 44 | 50 | 53
Fever (General disorders) | 16 | 26 | 31
Irritability (General disorders) | 56 | 62 | 70
Loss of appetite (General disorders) | 33 | 40 | 48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.